CLINICAL TRIAL: NCT01539356
Title: Hepcidin Levels in Preterm Infants Receiving Blood Transfusion and During Sepsis.
Brief Title: Hepcidin Levels in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0154-11-MMC
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2012-11

CONDITIONS: Preterm Infants; Anemia of Prematurity; Neonatal Sepsis
Keywords: Hepcidin; Preterm Infants; Anemia; Sepsis; Ferritin
MeSH Terms: conditions — Anemia; Neonatal Sepsis; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- preterm infants: preterm infants receiving blood transfusion
  preterm infants with neonatal sepsis.

SUMMARY:
A recently isolated peptide hormone, hepcidin, is thought to be the principal regulator of iron homeostasis. Hepcidin acts by limiting intestinal iron absorption and promoting iron retention in reticuloendothelial cells. The aims of this study were to determine serum hepcidin levels in preterm infants who receive blood transfusion and preterm infants having sepsis, in order to assess possible relationships between hepcidin and serum iron, serum ferritin,in iron load situations.

ELIGIBILITY:
Inclusion Criteria:

* Preterm < 38 weeks gestation
* Need of blood test for anemia or suspected sepsis

Exclusion Criteria:

* Major congenital anomalies
* Birth Asphyxia

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm < 38 weeks gestation Need of blood transfusion according to local Protocol. or signs and symptoms of sepsis
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Increase in Hepcidin levels by 30% | within 24-72 h

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Intensive Care Unit, Kfar Saba, Israel

REFERENCES:
- [Background] Muller KF, Lorenz L, Poets CF, Westerman M, Franz AR. Hepcidin concentrations in serum and urine correlate with iron homeostasis in preterm infants. J Pediatr. 2012 Jun;160(6):949-53.e2. doi: 10.1016/j.jpeds.2011.12.030. Epub 2012 Jan 28. PMID 22284565
- [Background] Yapakci E, Tarcan A, Celik B, Ozbek N, Gurakan B. Serum pro-hepcidin levels in term and preterm newborns with sepsis. Pediatr Int. 2009 Apr;51(2):289-92. doi: 10.1111/j.1442-200X.2008.02688.x. PMID 19405934